CLINICAL TRIAL: NCT00735033
Title: The Effects of the Swiss Ball on Patients With Hemiplegia Due to Cerebral Vascular Accident
Brief Title: The Effects of the Swiss Ball on Cerebral Vascular Accident
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fortaleza University (Other)
Purpose: Treatment
Other Study IDs: coetica-130/2004
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-05

CONDITIONS: Hemiplegia; Cerebrovascular Accident
Keywords: Physical therapy; Physical therapy modalities; Cerebral Vascular Accident (CVA)
MeSH Terms: conditions — Hemiplegia; Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Physiotherapy with Swiss Ball

SUMMARY:
The objective of this study was to investigate the effects of the Swiss ball on patients with hemiplegia due to CVA.

DETAILED DESCRIPTION:
The Cerebral Vascular Accident (CVA) is a neurological deficit, which may be transitory or definite, leading to motor, psychological and social alterations. It's the third cause of death in the industrialized world, of which 90% of the survivors have some residual deficit and 30% become disabled. The objective of this study was to investigate the effects of the Swiss ball on patients with hemiplegia due to CVA. An intervening and controlled study was conducted on 12 patients of both genders and over 50 years old with chronic hemiplegia, all undergoing treatment at the Beneficent Rehabilitation Association of Ceará. The patients in the experimental group (EG) underwent treatment with the Swiss ball added to conventional physical therapy and the control group (CG) went through conventional physiotherapy sessions. The treatment was done twice a week, consisting of 14 sessions altogether. The data were collected in an evaluation form at the beginning and at the end of the treatment. Most patients were found to be males; they had typical walking ability, tonus, and posture of chronic hemiplegia patients. The patients in the experimental group showed significantly greater muscular strength on the lower limbs than the control group (p < 0,05, Student t test), however, the same did not happen in the case of the other parameters, such as strength on the upper limbs, coordination, and balance. We can conclude that the treatment with the Swiss ball can promote increased strength, which will allow for a more efficient recovery in the studied population.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia due to CVA
* In physiotherapy treatment
* Acceptance in join the research

Exclusion Criteria:

* Less then 6 months of diagnostic

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult